CLINICAL TRIAL: NCT04728906
Title: Targeted-cell Therapy Using Epithelial Stem Cells and Patients' Cardiomyocytes Loaded in Amnion Bilayer to Regenerate Myocardial Infarction Post COVID-19 Complication
Brief Title: Heart Patch for Myocardial Infarction COVID-19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rumah Sakit Pusat Angkatan Darat Gatot Soebroto (Other)
Collaborators: Fakultas Kedokteran Universitas Indonesia (Other); RSUPN dr. Cipto Mangunkusumo (Unknown); Rumah Sakit Universitas Indonesia (Unknown); Pusat Jantung Nasional Harapan Kita (Unknown)
Responsible Party: Principal Investigator, Normalina Sandora, Normalina Sandora, MD, MSc, PhD, Rumah Sakit Pusat Angkatan Darat Gatot Soebroto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 120/KEPK-RSB/X/20
Record Dates: First submitted 2021-01-26; First posted 2021-01-28 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Myocardial Infarction; Heart Diseases
MeSH Terms: conditions — Myocardial Infarction; Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Heart patch + cardiomyocytes - hAESC (Experimental): Patients who undergo bypass (CABG) surgery are given heart patch in areas where grafting (bypass) is not feasible
  Interventions: Device: Heart patch seeded with autologous cardiomyocytes and amnion epithelial stem cells

INTERVENTIONS:
Device: Heart patch seeded with autologous cardiomyocytes and amnion epithelial stem cells — heart patch is seeded with patient's cardiomyocytes (taken from patient's heart waste tissue when undergoing bypass surgery) and stock amnion epithelial stem cells (HLA-DR negative to eliminate risk of rejection)

SUMMARY:
Myocardial infarction (MI), as one of the many complications of COVID-19, is one of the contributing patients of patients' death. This study attempts on developing an intervention of MI by regenerating damaged cardiomyocytes due to insufficiency of oxygen in cardiac muscles, triggered by an occlusion of coronary artery (MI). Heart patch developed from amnion bilayer seeded with amnion epithelial stem cells and patient's autologous cardiomyocytes is used as a therapy. Patients who undergo bypass (CABG) surgery are given heart patch, and then patients condition are observed by ECG, Echo, blood test, and radiology (technetium-99m)

ELIGIBILITY:
Inclusion Criteria:

* Aged 40 - 60 years old
* Ischemic burden >10% and ischemic gradients red-violet
* Ischemic area is not feasible to be grafted (bypass) due to other conditions such as diffusion and deep intramuscular vascularization
* Ejection fraction >30-35%
* Euro score <8

Exclusion Criteria:

* Scanning of Technetium-99 showed black colored ischemic area
* Patients undergoing other procedures other than bypass such as valve repair
* Chronic kidney failure
* Patients have went through several bypass surgeries prior
* Patients are still COVID-19 positive
* Immunocompromised patients

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Change of the ischemic burden (%) | Comparison from the imaging within 3 months before intervention, and after 6 months post treatment.
  Diagnosed by MRI
Change in the regional heart wall motion abnormality | Observation of the heart wall motion by 1 week before intervention and 4 - 12 - 24 weeks after intervention
  measured using Echocardiographic

SECONDARY OUTCOMES:
Change of the electrocardiographic wave | Observation of electrocardiogram records by 1 week before intervention and 4 - 12 - 24 weeks after intervention
  Measured using electrocardiogram
Change of the ejection fraction | Observation of the heart motion by 1 week before intervention and 4 - 12 - 24 weeks after intervention
  Measured using echocardiography

CONTACTS AND LOCATIONS:
Locations (3):
- Indonesia (3):
  - RSUPN dr. Cipto Mangunkusumo, Jakarta, DKI Jakarta
  - Rumah Sakit Universitas Indonesia, Depok, West Java
  - Pusat Jantung Nasional Harapan Kita, Jakarta

IPD SHARING:
Plan to Share IPD: No